CLINICAL TRIAL: NCT03547557
Title: MR Guided Focused Ultrasound Surgery in the Treatment of Pain Resulting From Metastatic Bone Tumors With the ExAblate 2000 Strappable System
Brief Title: MR Guided Focused Ultrasound Surgery in the Treatment of Pain From Bone Tumors w/ the ExAblate 2000 Strappable System
Acronym: BM005
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BM005
Record Dates: First submitted 2012-09-13; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Bone Metastases
Keywords: Bone Tumors
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ExAblate MRgFUS (Experimental)
  Interventions: Device: Exablate 2000 strappable system

INTERVENTIONS:
Device: Exablate 2000 strappable system

SUMMARY:
A Feasibility Study To Evaluate the Safety and initial Effectiveness of MR guided Focused Ultrasound Surgery in the Treatment of pain resulting from Metastatic Bone Tumors with the ExAblate 2000 strappable system.

DETAILED DESCRIPTION:
Bone is the third most common organ involved by metastatic disease behind lung and liver. In breast cancer, bone is the second most common site of metastatic spread, and 90% of patients dying of breast cancer have bone metastasis. Breast and prostate cancer metastasize to bone most frequently, which reflects the high incidence of both of these tumors, as well as their prolonged clinical courses.

Post cancer survival has increased with improvement in early detection and treatments. As a consequence, the number of patients developing metastatic bone disease during their lifetime has also increased. Patients with bone metastasis from breast cancer have an average 2-year survival from the time of presentation with their first bone lesion. In patients who die from breast, prostate, and lung cancer, autopsy studies have shown that up to 85% have evidence of bone metastases at the time of death.

Current treatments for patients with bone metastases are primarily palliative and include localized therapies (radiation and surgery), systemic therapies (chemotherapy, hormonal therapy, radiopharmaceutical, and bisphosphonates), and analgesics (opioids and non-steroidal anti-inflammatory drugs). Recently, radiofrequency ablation has been tested as a treatment option for bone metastases. The main goals of these treatments are improvement of quality of life and functional level. These goals can be further described: 1) Pain relief, 2) Preservation and restoration of function, 3) Local tumor control, 4) Skeletal stabilization.

The study hypothesis is that treatment with the MRgFUS, which is delivered by a strappable transducer, is a safe and potentially effective non-invasive treatment for metastatic bone tumors with a low incidence of co-morbidity. Based on the results of this study the Sponsor will initiate a larger study in an attempt to obtain regulatory approval for the treatment of metastatic bone tumors as an indication for the MRgFUS ExAblate strappable system.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 and older
2. Patients who are able and willing to give written consent and are able to attend all study visits
3. Patients with histologically or cytologically confirmed malignant disease with a bone lesion that appears to be metastatic disease by clinical and or imaging techniques
4. Patients with persistent pain from at least one site of bone metastases and are able to distinguish the pain from other painful sites oPatient with localized VAS pain score ≥ 4, at the target tumor oIn case of patients with more than one painful site, VAS pain score at the target site should exceed VAS pain score at any other site by at least two units.
5. Targeted tumor(s) are ExAblate device accessible and are located in ribs, extremities (excluding joints), pelvis, shoulders and in the posterior aspects of the following spinal vertebra: Lumbar vertebra (L3 - L5), Sacral vertebra (S1 - S5)
6. Targeted tumor(s) size is smaller than 8 cm in diameter on bone surface
7. Patient whose lesion is on bone and is ≥ 10-mm from the skin.
8. Tumor(s) clearly visible by non-contrast MRI
9. Able to communicate sensations during the MRgFUS ExAblate treatment
10. KPS ≥60 (See "Definitions" below)
11. At least 2 weeks since chemotherapy
12. At least 1 month since radiation therapy

Exclusion Criteria:

1. Diffuse skeletal tumoral spread as evaluated by imaging.
2. Patients who need pre-treatment surgical stabilization of the affected bony structure.
3. Targeted tumor is in impending fracture
4. Patients with unstable cardiac status including:

   * Unstable angina pectoris on medication oPatients with documented myocardial infarction within six months of protocol entry oCongestive heart failure requiring medication (other than diuretic) oPatients on anti-arrhythmic drugs
5. Severe hypertension (diastolic BP > 100 on medication)
6. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations; weight >110 kg, etc.
7. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist)
8. Extensive scarring in an area in the path of energy planned passage to the treatment area
9. Severe cerebrovascular disease (multiple CVA or CVA within 6 months)
10. Patients on anti-coagulation therapy or those with an underlying bleeding disorder
11. Severely abnormal coagulation (INR>1.5)the upper limit
12. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 2 hrs.)
13. Patients with life expectancy < 6-Months
14. Patients with surgical stabilization of tumor site with metallic hardware
15. Lesion is less then 5mm from a nerve.
16. Pregnant or lactating women
17. Patients that are currently participating or have participated in another clinical trial in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | Within 3 months of treatment
  adverse event incidence and severity
Change in pain Numerical Rating Scale (NRS) from pre-treatment to post treatment | 3 months post treatment
  NRS scale 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Prof. R. Catane, Principal Investigator — Sheba Medical Center-Oncology Division
Locations (1):
- Sheba Medical Center Oncology Department, Tel Litwinsky, Israel

REFERENCES:
- See also: Sponsor's Web Page — http://www.insightec.com